CLINICAL TRIAL: NCT04087967
Title: A Phase 3, Randomized, Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of Decitabine Combined With HAAG Regimen in Newly Diagnosed Acute Myeloid Leukemia Patients Younger Than 60 Years
Brief Title: Study of DAC Combined With HAAG Regimen in Newly Diagnosed Younger AML Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other); Changzhou No.2 People's Hospital (Other); The First People's Hospital of Lianyungang (Other); Jingjiang People's Hospital (Other); Zhangjiagang First People's Hospital (Other); The Second People's Hospital of Huai'an (Other); The Third People's Hospital of Kunshan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAC-HAAG-01
Record Dates: First submitted 2019-09-08; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Acute Myeloid Leukemia; Induction Chemotherapy
Keywords: Decitabine; HAAG; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Idarubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine combined with HAAG (Experimental): This cohort will determine the safety and efficacy of decitabine combined with HAAG regimen in the newly diagnosed AML patients younger than 60.
  Interventions: Drug: Decitabine plus HAAG regimen
- IA Regimen (Active Comparator): This cohort will determine the safety and efficacy of decitabine combined with HAAG regimen in the newly diagnosed AML patients younger than 60.
  Interventions: Drug: Idarubicine plus Cytarabine regimen

INTERVENTIONS:
Drug: Decitabine plus HAAG regimen — Decitabine:20mg/m2/d,d1~5, intravenous infusion; Homoharringtonine:1mg/d,d3~16,intravenous infusion; Aclarubicin:10mg/d, d3~d10, intravenous infusion; Cytarabine:10mg/m2,q12h,d3-16, subcutaneous injection;
  Granulocyte colony-stimulating factor (G-CSF):
  50-300μg/d (when WBC counts are less than 20×10^9/L ),subcutaneous injection;
  Arms: Decitabine combined with HAAG
Drug: Idarubicine plus Cytarabine regimen — Idarubicine :12mg/m2, d1-3, intravenous infusion; Cytarabine :100mg/m2, d1-7, 24-hours continuous intravenous infusion
  Arms: IA Regimen

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of DAC combined with HAAG regimen in the induction treatment of newly diagnosed AML patients younger than 60 years.

DETAILED DESCRIPTION:
This is a phase 3, randomized, controlled, multi-center study in newly diagnosed AML patients younger than 60. The patients will be randomized to receive either DAC combined with HAAG or IA regimen in the induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML according to the WHO (2016) classification of acute myeloid leukemia.
2. Age 18-59.
3. ECOG score: 0-2.
4. Treatment related or secondary AML.
5. No history of previous chemotherapy or target therapy.
6. Provide informed consent.

Exclusion Criteria:

1. Patients are pregnant or lactating.
2. Patients have acute promylocytic leukemia or chronic myeloid leukemia in blast crisis.
3. Patients with another malignant disease.
4. Patients with uncontrolled active infection.
5. Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
6. Patients with aspartate aminotransferase or glutamic-pyruvic transaminase > 3x upper limit of normal or bilirubin > 2.0 mg/dL.
7. Patients with creatinine clearance rate < 50ml/min.
8. Patients with active hepatitis B or hepatitis C infection.
9. Patients with HIV infection.
10. Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Day 28-35 of induction course
  ORR includes complete response (CR), CRi and PR. CR was defined as < 5% bone marrow blasts in an aspirate with spicules, no blasts with Auer rods or persistence of extramedullary disease, and independent of transfusions; CRi: was defined as<5% bone marrow blasts, either ANC<1×10^9/L or platelets<100×10^9/L, transfusion independence but with persistence of cytopenia; PR was defined as decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow aspirate and the normalization of blood counts.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  time from randomization to death from any cause
Leukemia-free survival (LFS) | 3 years
  time from randomization to the first relapse or death
Cumulative incidence of relapse(CIR) | 3 years
  time from achievement of a remmission to the first relapse
Number of adverse events | 2 years
  adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China